CLINICAL TRIAL: NCT07362823
Title: A Study on the Efficacy of the Metaverse Lifestyle Health Education Model Based on the Transtheoretical Model for Improving Quality of Life and Modifying Lifestyle in Colorectal Cancer Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qu Shen (Other)
Responsible Party: Sponsor-Investigator, Qu Shen, Associate Professor, Xiamen University
Organization: Xiamen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: XDYX202510K58
Record Dates: First submitted 2025-12-27; First posted 2026-01-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Neoplasms; Cancer Survivors
Keywords: Colorectal Neoplasms; Cancer Survivors; Transtheoretical Model (TTM); Metaverse; Lifestyle Intervention; Health Education; Quality of Life; Self-Efficacy; Health Behavior; Multicenter Randomized Controlled Trial
MeSH Terms: conditions — Colorectal Neoplasms; Health Education; Health Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TTM-Based Metaverse Lifestyle Health Education Arm (Experimental): Administer TTM-phased lifestyle health education via metaverse platform (including health courses, immersive interactions, peer communities) and WeChat group check-in/medical Q&A. Assess indicators at baseline, 1-month, 3-month post-intervention.
  Interventions: Behavioral: TTM-Based Metaverse Lifestyle Health Education
- Routine Colorectal Cancer Postoperative Health Education Arm (No Intervention): Provide paper-based postoperative rehabilitation manual and verbal lifestyle guidance; conduct routine telephone/outpatient follow-up per hospital protocol. Assess indicators at the same time points as the intervention arm.

INTERVENTIONS:
Behavioral: TTM-Based Metaverse Lifestyle Health Education — A three-month, stage-stratified behavioral intervention targeting colorectal cancer postoperative survivors, developed in alignment with the five stages of the Transtheoretical Model (TTM): pre-contemplation, contemplation, preparation, action, and maintenance. The intervention encompasses lifestyle modification modules (encompassing dietary guidance, physical activity protocols, and stress management) delivered via a metaverse platform-including didactic materials, immersive interactive modules, health behavior challenges, and peer support communities (20-30 minutes daily). It is supplemented by daily check-in prompts via WeChat groups and real-time clinical consultation from the research team. This intervention is designed to facilitate the adoption of health-promoting behaviors and enhance health-related quality of life among participants.
  Other Names: TTM-Metaverse Health Education
  Arms: TTM-Based Metaverse Lifestyle Health Education Arm

SUMMARY:
Colorectal cancer is a globally prevalent malignant tumor. Postoperative patients often face physical discomfort, psychological stress, and lack of healthy lifestyles. However, traditional health education models have limitations such as insufficient targeting and poor interactivity, making it difficult to meet their needs for full-cycle health management. This study is a multicenter randomized controlled trial, which plans to enroll 174 patients aged 18 years and above who have undergone radical resection for colorectal cancer, and randomly divide them into an experimental group and a control group at a ratio of 1:1. The experimental group will receive Transtheoretical Model (TTM)-based metaverse lifestyle health education (including phased course learning, metaverse immersive interaction, and WeChat group check-in supervision) with an intervention cycle of 1 months and follow-up until 3 months after the intervention; the control group will only receive routine paper-based education and outpatient follow-up. The study aims to verify the improvement effect of this metaverse intervention model on the quality of life and healthy lifestyle of colorectal cancer survivors, and explore its role in improving patients' self-efficacy, so as to provide empirical evidence for optimizing long-term health management programs for cancer survivors.

DETAILED DESCRIPTION:
1. Study Background Colorectal cancer ranks 2nd in incidence and 4th in mortality among malignant tumors in China, with 517,000 new cases and 240,000 deaths in 2022, and the number of patients is expected to increase to 910,000 by 2040. Surgical and other treatment methods have prolonged patients' survival, transforming the disease into a chronic condition requiring long-term management. However, postoperative patients generally experience physical symptoms such as pain and gastrointestinal disorders, as well as psychological problems such as fear of recurrence and anxiety, and have low compliance with healthy lifestyle behaviors such as balanced diet and regular exercise. Traditional health education mainly relies on paper manuals and verbal guidance, lacking phased behavioral interventions and continuous interactive support, which cannot effectively promote the development of long-term healthy behaviors in patients.

   The Transtheoretical Model (TTM) divides behavior change into 5 stages (pre-contemplation, contemplation, preparation, action, maintenance) and can provide targeted behavioral intervention strategies; metaverse technology has the advantages of immersion and high interactivity, which can break the temporal and spatial limitations of traditional education. This study integrates TTM theory, lifestyle medicine (including six pillars such as diet, exercise, and stress management) and metaverse technology to build a new health education model, aiming to address the core pain points of health management for colorectal cancer survivors.
2. Study Design

   This is a prospective multicenter randomized controlled trial conducted in 3 Grade A tertiary hospitals: The First Affiliated Hospital of Xiamen University, Zhongshan Hospital Affiliated to Xiamen University, and Xiang'an Hospital Affiliated to Xiamen University. The study is divided into 3 phases:

   2.1 Theoretical Construction Phase: Develop phased lifestyle health education courses based on TTM through literature research and expert consultation, and complete the functional adaptation of the metaverse platform (including modules such as graphic and text education, course learning, health challenges, and patient communities); 2.2 Intervention Implementation Phase: After signing the informed consent form, eligible patients are randomly grouped by tumor stage and age through the central randomization system (REDCap platform). The experimental group receives 3-month metaverse intervention (3 days for pre-contemplation stage, 4 days for contemplation stage, 7 days for preparation stage, 14 days for action stage, 14 days for maintenance stage, with a daily intervention duration of 20-30 minutes), and completes daily check-ins and medical Q&A through WeChat groups; the control group receives routine health education (distribute the Postoperative Rehabilitation Manual for Colorectal Cancer and complete postoperative follow-up according to hospital procedures); 2.3 Effect Evaluation Phase: Collect patients' quality of life (FACT-C scale), healthy lifestyle (HPLP II scale), self-efficacy (SUPPH scale), and physiological indicators such as BMI and CEA before intervention (T0), 1 month after intervention (T1), and 3 months after intervention (T2). Meanwhile, record the usage compliance of the metaverse platform and adverse events.
3. Study Endpoints 3.1 Primary Endpoints: Changes in standardized scores of the FACT-C scale and scores of the HPLP II scale in patients at 3 months after intervention (T2) compared with baseline (T0); 3.2 Secondary Endpoints: Changes in SUPPH scale scores, progress of behavior change stages, improvement of physiological indicators, platform usage compliance and satisfaction of patients during T0-T2; 3.3 Safety Endpoints: Incidence and severity of adverse events (such as exercise-related muscle soreness and platform operation discomfort) during the intervention period.
4. Quality Control The research team will conduct a unified baseline assessment of enrolled patients, and intervention personnel will take up their posts after passing GCP and platform operation training and assessment; double independent data entry is adopted, and missing values are handled by multiple imputation; meanwhile, a monitoring group is established to verify data from each center every 2 months to ensure the accuracy and completeness of research data.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with first diagnosed colorectal cancer who have undergone radical surgical treatment
2. Aged ≥18 years old and non-pregnant
3. Have basic communication, reading and comprehension abilities, and can proficiently use smartphones and WeChat
4. Voluntarily sign the informed consent form and promise to cooperate in completing all interventions and follow-up assessments

Exclusion Criteria:

1. Patients with other types of malignant tumors
2. Patients with incompletely resected tumors or distant metastases
3. Patients with dysfunction of important organs such as heart, liver and kidney, or with unstable/rapidly deteriorating conditions
4. Patients with severe cognitive impairment who cannot communicate normally and cooperate with the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Health-Related Quality of Life Assessed by the Functional Assessment of Cancer Therapy-Colorectal (FACT-C) Scale | Baseline (T0), 1 month after intervention (T1), 3 months after intervention (T2)
  The FACT-C scale, a colorectal cancer-specific validated instrument, comprises 36 items across 5 domains (physical, social/family, emotional, functional well-being, and colorectal cancer-specific subscale). Scores are standardized to a 0-100 range, with higher scores indicating better quality of life. The outcome measures the change in standardized scores from baseline to 1 mouth and 3 months post-intervention.
Improvement in Health-Promoting Behaviors Assessed by the Health-Promoting Lifestyle Profile II (HPLP II) Scale | Baseline (T0), 1 month after intervention (T1), 3 months after intervention (T2)
  The HPLP II scale includes 52 items across 6 domains (self-actualization, health responsibility, physical activity, nutrition, interpersonal support, stress management). Scores range from 52 to 208, with higher scores reflecting more consistent health-promoting behaviors. The outcome measures the change in total scores from baseline to 1 month and 3 months post-intervention.

SECONDARY OUTCOMES:
Change in Self-Efficacy Assessed by the Strategies Used by People to Promote Health (SUPPH) Scale | Baseline (T0), 1 month after intervention (T1), 3 months after intervention (T2)
  The SUPPH scale is a validated instrument for cancer patients, consisting of 28 items across 3 domains (positive attitude, self-stress reduction, self-decision-making). Scores range from 28 to 140, with higher scores indicating stronger self-efficacy. The outcome measures the change in total scores at 1-month and 3-month post-intervention compared with baseline.
Progression of Health Behavior Change Stages Assessed by the Transtheoretical Model (TTM) Stage Scale | Baseline (T0), 1 month after intervention (T1), 3 months after intervention (T2)
  The TTM Stage Scale classifies behavior change into 5 stages (pre-contemplation, contemplation, preparation, action, maintenance). The outcome evaluates the progression of participants' stages (defined as advancing at least one stage) at 1-month and 3-month post-intervention relative to baseline.
Change in BMI | Baseline (T0), 1 month after intervention (T1), 3 months after intervention (T2)
  Key physiological indicators include body mass index (BMI). The investigators collect BMI data via hospital laboratory tests to assess metabolic and tumor-related health status changes.
Change in CEA | Baseline (T0), 1 month after intervention (T1), 3 months after intervention (T2)
  Carcinoembryonic antigen (CEA) is a key physiological indicator. The investigators collect the data via hospital laboratory tests.
Change in Blood Glucose | Baseline (T0), 1 month after intervention (T1), 3 months after intervention (T2)
  The investigators collect the data of fasting blood glucose via hospital laboratory tests to assess metabolic and tumor-related health status changes.
Change in Blood Lipids | Baseline (T0), 1 month after intervention (T1), 3 months after intervention (T2)
  The investigators collect the data of total cholesterol, triglycerides, low-density lipoprotein (LDL), and high-density lipoprotein (HDL) via hospital laboratory tests to assess metabolic and tumor-related health status changes.
Intervention Adherence Rate of Metaverse Platform Usage | Weekly during the 3-month intervention period; summarized at 3 months after intervention (T2)
  Adherence is defined as the percentage of actual completed intervention tasks (including daily metaverse platform usage and course learning) relative to the required tasks. A rate ≥70% is classified as high adherence.
Participant Satisfaction with the Metaverse Health Education Platform | 1 month after intervention (T1), 3 months after intervention (T2)
  Assessed by a validated self-designed questionnaire (5-point Likert scale) covering platform functionality, course content relevance, interactive experience, and perceived intervention benefits. Higher scores indicate greater satisfaction.